CLINICAL TRIAL: NCT04058418
Title: Impact of Familial Cancer Specialist Recommendation on Chemoprevention Prescribing for Familial Breast Cancer (FBC) Risk in Primary Care: Short Survey and Interrupted Time Series Analysis
Brief Title: Specialist Recommendation on FBC (Familial Breast Cancer) Chemoprevention Prescribing
Acronym: FBC
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 19049
Record Dates: First submitted 2019-06-12; First posted 2019-08-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Familial Breast Cancer
MeSH Terms: conditions — Breast Cancer, Familial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Familial breast cancer risk assessment services in England: All familial breast cancer risk assessment services in England
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Completion of a short survey.

SUMMARY:
Some women are more likely to get breast cancer as it runs in their family, they are at risk of familial breast cancer. There are medications, called chemoprevention, which may lower their risk of developing breast cancer by a third. However chemoprevention can also cause serious side effects, like womb cancer and blood clots. This makes decision to start them difficult. Researchers found that not all women who can have these medications are on them.

The investigators want to ask familial breast cancer specialists whether they recommend general practitioners (GP) to prescribe chemoprevention, by sending them a short survey. These specialists look after women where breast cancer runs in the family. The specialists assess a women's chance of getting breast cancer and advice those with increased risk what can be done to prevent breast cancer.

The investigators will then look at whether specialist recommendation makes a difference to whether GPs prescribe chemoprevention medication. This will be done by linking the specialists' survey response to information on GP prescribing that the government regularly publishes. This may help the investigators understand why chemoprevention is not used as often as it potentially can be.

DETAILED DESCRIPTION:
Phase I: Short survey of lead clinicians of familial cancer services, descriptive analysis of recommendations by areas of the country

Phase II: Prescribing data analysis (using OpenPrescribing) comprising:

1. t-test to compare the chemoprevention prescribing rate in general practices where chemoprevention is recommended versus not recommended;
2. interrupted times series analysis to assess the change in the chemoprevention prescribing after recommendation from specialist compared with changes occurring in practices where chemoprevention is not recommended and
3. panel regression across all practices, in order to distinguish the relative impacts of national versus local recommendation, and the change over time.

ELIGIBILITY:
Inclusion Criteria:

* Lead clinicians of NHS familial cancer services across England
* Standard general practices (classed as type 4 by NHS Digital, to exclude walk-in centres, prisons, care homes, etc.) with prescribing data for chemoprevention available on OpenPrescribing

Exclusion Criteria:

* General practices with less than 10 female patients aged 35 to 44 registered
* General practices which cannot be linked to any familial cancer service from survey responses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: NHS familial cancer services and general practices in England
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of specialist service that recommends chemoprevention prescribing by areas in England | 2019
  Proportion of specialist service that recommends chemoprevention prescribing by areas in England, measured using survey questionnaire
Chemoprevention medication prescribing rates in primary care by area in England | post specialist recommendation over 24 months
  2.1. The chemoprevention prescribing rate in general practices where chemoprevention is recommended versus not recommended. The rate will be measured as the number of average daily quantities (ADQs) of chemoprevention prescribed per 1000 registered female patients aged between 35 and 74 per practice. For our primary outcome we will measure only tamoxifen items, and assess other therapies used in chemoprevention in supplementary analyses.
  2.2. The change in chemoprevention prescribing rate (described in outcome 2.1) in general practices after recommendation from local specialist, compared with changes occurring in practices where chemoprevention is not recommended.
  2.3. The relative change in the chemoprevention prescribing rate (described in outcome 2.1) in general practice in response to local recommendation, compared with change occurring in response to national recommendation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Prescribing analysis code and raw data (of publicly available, anonymised, primary care prescribing data) will be made freely available alongside publication of results.

REFERENCES:
- [Background] Curtis HJ, Walker AJ, Goldacre B. Impact of NICE guidance on tamoxifen prescribing in England 2011-2017: an interrupted time series analysis. Br J Cancer. 2018 May;118(9):1268-1275. doi: 10.1038/s41416-018-0065-2. Epub 2018 Apr 23. PMID 29681615
- [Background] Qureshi N, O'Flynn N, Evans G. Dealing with family history of breast cancer: something new, something old. Br J Gen Pract. 2014 Jan;64(618):6-7. doi: 10.3399/bjgp14X676267. No abstract available. PMID 24567549